CLINICAL TRIAL: NCT03733171
Title: Role of Platelet Rich Plasma in the Treatment of Actively Bleeding Peptic Ulcer
Brief Title: Platelet Rich Plasma in Bleeding Peptic Ulcer
Acronym: PRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Hanafy, Assistant professor of medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4940
Record Dates: First submitted 2018-11-05; First posted 2018-11-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Bleeding Ulcer
Keywords: platelet rich plasma
MeSH Terms: interventions — Hemostasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma (Active Comparator): endoscopic injection of PRP
  Interventions: Drug: PLATELET RICH PLASMA
- CONTROL GROUP (Placebo Comparator): diluted epinephrine
  Interventions: Drug: diluted epinephrine; Device: hemoclips

INTERVENTIONS:
Drug: PLATELET RICH PLASMA — PRP was injected in 1-2 ml by multiple injections into and circumferentially around the ulcer until bleeding stopped using a 25-G retractable, standard sclerotherapy needle
  Other Names: PRP
  Arms: Platelet rich plasma
Drug: diluted epinephrine — diluted epinephrine was injected in 1-2 ml by multiple injections into and circumferentially around the ulcer until bleeding stopped using a 25-G retractable, standard sclerotherapy needle
  Other Names: Hemostasis
  Arms: CONTROL GROUP
Device: hemoclips — diluted epinephrine was injected followed by application of hemoclips
  Other Names: mechanical hemostasis
  Arms: CONTROL GROUP

SUMMARY:
The most common cause of acute upper gastrointestinal bleeding (UGIB) is non-variceal, where peptic ulcer bleeding (PUB) remains the single most common cause, accounting for 25% to 67% of the causes of non-variceal upper gastrointestinal bleeding (NVUGIB).

Despite major advances in diagnostic and therapeutic tools, PUB remains a significant problem and an important cause of morbidity and mortality. Given the imperative therapeutic role of endoscopic management in achieving hemostasis in NVUGIB, new modalities to improve the current treatment strategies continue to be developed.

Platelet-rich plasma (PRP) is a widely used throughout many fields of medicine for improving tissue regeneration. PRP contains a higher concentration of platelets than whole blood, and represents a pool of many growth-factors.

DETAILED DESCRIPTION:
All patients were subjected to full history taking, complete clinical examination, laboratory investigations (complete blood count, liver and kidney function tests, coagulation profile), ECG and Upper GI endoscopy was performed within 24 hours of hospital admission after initial resuscitation of patients including blood transfusion if HB level ≤ 7g ∕ L.

Stigmata of recent hemorrhage was defined according to the Forrest (F) classification (FIa- spurting hemorrhage, FIb- oozing hemorrhage, FIIa- non-bleeding visible vessel, FIIb- adherent clot, FIIc- flat pigmented spot and FIII- clean base ulcer).The size of an ulcer was classified as < 2 cm or ≥ 2cm.

* PRP or diluted epinephrine were injected in 1-2 ml by multiple injections into and circumferentially around the ulcer until bleeding stopped using a 25-G retractable, standard sclerotherapy needle.
* Group I was subjected to multiple injection of PRP (each 1-2 ml), while group II was subjected to epinephrine injections (each 1-2 ml of a 1:10.000 solution of epinephrine) .
* Hemostasis was achieved if bleeding stopped for at least 3 min of observation. Immediately after the endoscopic hemostasis, PPIs were infused at a standard regimen (40 mg bolus of PPI once daily for 72 h) or at a high-dose regimen (loading dose of 80 mg on the first day followed by continuous infusion of 8 mg/h for 72 h), after the initial 72 h, patients were switched to oral PPIs (20 mg twice daily) until discharge .

PRP preparation method

Under complete aseptic conditions the blood was drawn with the addition of anticoagulant such as citrate dextrose A to prevent platelet activation prior to its use.

1.30-60 cc of patients' blood drawn at the time of treatment by venipuncture in acid citrate dextrose (acts as an anticoagulant) tubes 2. Do not chill the blood. 3. Centrifuge the blood using a 'soft' spin (1st centrifugation). 4. Transfer the supernatant plasma containing platelets into another sterile tube (without anticoagulant).

5. Centrifuge tube at a higher speed (a hard spin) to obtain a platelet concentrate (2nd centrifugation).

6. The lower 1/3rd is PRP and upper 2/3rd is platelet-poor plasma (PPP). At the bottom of the tube, platelet pellets are formed.

7. Remove PPP and suspend the platelet pellets in a minimum quantity of plasma (2-4 mL) by gently shaking the tube.

8.Thrombin (dose) was added to activate PRP

ELIGIBILITY:
Inclusion Criteria:

* Patients who have a peptic ulcer with either actively bleeding or a non-bleeding visible vessel
* initial hemoglobin concentration of < 10 g/dL

Exclusion Criteria:

* Patients with non-PUB, coagulopathy, bleeding disorders, anticoagulant therapy, cardiopulmonary compromise, hypertension, ischemic heart disease, arrhythmia, and patients who refused to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
bleeding | 3 months
  control of peptic ulcer bleeding

SECONDARY OUTCOMES:
improved iron indices | 3 months
  imroved complete blood count element

CONTACTS AND LOCATIONS:
Overall Officials: WASEEM SELEEM, MD, Principal Investigator — zagazig university hospital
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

REFERENCES:
- [Derived] Seleem WM, Hanafy AS. The Additive Effect of Platelet-Rich Plasma in the Treatment of Actively Bleeding Peptic Ulcer. Clin Endosc. 2021 Nov;54(6):864-871. doi: 10.5946/ce.2021.004. Epub 2021 May 25. PMID 34030430